CLINICAL TRIAL: NCT01766817
Title: Safety and Efficacy of a Lysophosphatidic Acid Receptor Antagonist in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM136-003
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: BMS 986020, 600 mg. once daily (Experimental): BMS-986020, 600 mg tablets, by mouth, once daily, 26 weeks
  Interventions: Drug: BMS-986020
- Arm 2: BMS-986020, 600 mg twice daily (Experimental): BMS-986020, 600 mg tablets, by mouth, twice daily, 26 weeks
  Interventions: Drug: BMS-986020
- Arm 3: Placebo matching with BMS-986020 (Placebo Comparator): Placebo, 0 mg tablets, by mouth, twice daily, 26 weeks
  Interventions: Drug: Placebo matching with BMS-986020

INTERVENTIONS:
Drug: BMS-986020
  Arms: Arm 1: BMS 986020, 600 mg. once daily; Arm 2: BMS-986020, 600 mg twice daily
Drug: Placebo matching with BMS-986020
  Arms: Arm 3: Placebo matching with BMS-986020

SUMMARY:
The purpose of this study is to determine if study drug (BMS-986020) dose of 600 mg once daily or 600 mg twice daily for 26 weeks compared with placebo will reduce the decline in forced vital capacity (FVC) and will be well tolerated in subjects with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 40 and 90 years, inclusive, at randomization.
* Have clinical symptoms consistent with IPF.
* Have first received a diagnosis of IPF less than 6 years before randomization. The date of diagnosis is defined as the date of the first available imaging or surgical lung biopsy consistent with IPF/UIP.
* Have a diagnosis of usual interstitial pulmonary fibrosis (UIP) or IPF by HRCT or surgical lung biopsy (SLB).
* Extent of fibrotic changes (honeycombing, reticular changes) greater than the extent of emphysema on HRCT scan.
* Have no features supporting an alternative diagnosis on transbronchial biopsy, BAL, or SLB, if performed.
* Have percent predicted post-bronchodilator FVC between 45% and 90%, inclusive, at screening.
* Have a change in post-bronchodilator FVC (measured in liters) between screening and day 1 that is less than a 10% relative difference, calculated as: the absolute value of 100% * (screening FVC (L) - day 1 FVC (L)) / screening FVC (L).
* Have carbon monoxide diffusing capacity (DLCO) between 30% and 80% (adjusted for hemoglobin and altitude), inclusive, at screening.
* Have no evidence of improvement in measures of IPF disease severity over the preceding year, in the investigator's opinion.
* Be able to walk 150 meters or more at screening.
* Demonstrate an exertional decrease in oxygen saturation of 2 percentage points or greater at screening (may be performed with supplemental oxygen titrating to keep oxygen saturation levels >88%).
* Are able to understand and sign a written informed consent form.
* Are able to understand the importance of adherence to study treatment and the study protocol and are willing to comply with all study requirements, including the concomitant medication restrictions, throughout the study.
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must use acceptable method(s) of contraception. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is less than 24 hours, contraception should be continued for a period of 30 days after the last dose of investigational product.

  1. Women must have a negative urine pregnancy test within 24 hours prior to the start of investigational product.
  2. Women must not be breastfeeding.
  3. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is less than 24 hours, contraception should be continued for a period of 90 days after the last dose of investigational product.
  4. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception.

Exclusion Criteria:

Target Disease Exclusions

1. Has significant clinical worsening of IPF between screening and day 1 (during the screening process), in the opinion of the investigator.
2. Has forced expiratory volume in 1 second (FEV1)/FVC ratio less than 0.8 after administration of bronchodilator at screening.
3. Has bronchodilator response, defined by an absolute increase of 12% or greater and an increase of 200 mL in FEV1 or FVC or both after bronchodilator use compared with the values before bronchodilator use at screening.

Medical History and Concurrent Diseases

1. Has a history of clinically significant environmental exposure known to cause pulmonary fibrosis, including, but not limited to, drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds.
2. Has a known explanation for interstitial lung disease, including, but not limited to, radiation, drug toxicity, sarcoidosis, hypersensitivity, pneumonitis, bronchiolitis, obliterans, organizing pneumonia, human immunodeficiency virus (HIV), viral hepatitis, and cancer.
3. Has a clinical diagnosis of any connective tissue disease, including, but not limited to, scleroderma, polymyositis/dermatomyositis, systemic lupus erythematosus, rheumatoid arthritis, and undifferentiated connective tissue disease.
4. Currently has clinically significant asthma or chronic obstructive pulmonary disease.
5. Has clinical evidence of active infection, including, but not limited to, bronchitis, pneumonia, sinusitis, urinary tract infection, and cellulitis.
6. Has any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 2 years. This does not include minor surgical procedures for localized cancer (e.g., basal cell carcinoma).
7. Has any condition other than IPF that, in the opinion of the investigator, is likely to result in the death of the subject within the next 2 years.
8. Has a history of end-stage liver disease.
9. Has a history of end-stage renal disease requiring dialysis.
10. Has a history of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous 6 months, including, but not limited to, the following: i. Unstable angina pectoris or myocardial infarction ii. Congestive heart failure requiring hospitalization iii. Uncontrolled clinically significant arrhythmias
11. Has any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of BMS-986020.
12. Has a history of alcohol or substance abuse in the past 2 years.
13. Has a family or personal history of long QT syndrome and/or Torsades de Pointes (polymorphic ventricular tachycardia).
14. Has used any of the excluded medications per Appendix 1 of the Protocol, which includes, but is not limited to:

    * current treatment with pirfenidone or nintedanib
    * use of over-the-counter medications and herbal preparations, within 4 weeks before study drug administration except those medications cleared by the BMS medical monitor
    * For subjects taking statins, there are restrictions on the maximum allowable doses for statins listed below. If subjects are currently taking statins and their doses are higher than those mentioned below, please reduce the dose to the maximum allowable dose.

Additionally, if subjects are on statins and ready to start dosing, these subjects should limit statin doses by maximal allowable dose or lower for at least 5 days prior to the first BMS-986020 dosing. Shorter durations may be considered in select cases after discussion with the medical monitor.

Maximum allowable dose for statins:

* Simvastatin 20 mg QD
* Pitavastatin 2 mg QD
* Atorvastatin 40 mg QD
* Pravastatin 40 mg QD
* Rosuvastatin 20 mg QD
* Lovastatin 40 mg QD
* Fluvastatin 40 mg QD
* Prednisone is allowed up to a maximum of 15 mg po daily
* Pirfenidone or nintedanib dosing for a maximum of 3 months in the prior 12 months is permitted with a 4 week washout period prior to dosing with BMS-986020.

Physical and Laboratory Test Findings

1. Has any of the following liver-function test criteria above the specified limits: total bilirubin >1.5 x ULN, excluding subjects with Gilbert's syndrome; aspartate or alanine aminotransferase (AST/SGOT or ALT/SGPT) greater than 3 x ULN; alkaline phosphatase greater than 2.5 x ULN.
2. Has creatinine clearance less than 30 mL/minute, calculated using the Cockcroft-Gault formula.
3. Has ECG result with a QT interval by Fridericia's correction (QTcF) of 500 msec or greater or an uncorrected QT of 500 msec or greater at screening. Note: For subjects with a machine read QT interval of >500 msec, if their heart rate is > 100 bpm, the machine read QT interval (either corrected or not) may not be accurate. If the investigator is uncertain about the QT abnormality, it is recommended that ECGs be over-read by a cardiologist. The manually read QT interval by a cardiologist should be used for assessment of eligibility whenever possible.

Allergies and Adverse Drug Reaction Has had prior use of BMS-986020 or has known hypersensitivity to any of the components of study treatment.

Other Exclusion Criteria

1. Is not a suitable candidate for enrollment or is unlikely to comply with the requirements of this study, in the opinion of the investigator.
2. Has smoked cigarettes within 4 weeks or screening or is unwilling to avoid tobacco products throughout the study.
3. Is expected to receive a lung transplant within 1 year from randomization or, for subjects at sites in the United States, is on a lung-transplant waiting list at screening.
4. Prisoners or subjects who are involuntarily incarcerated.
5. Subjects who are compulsorily detained for treatment either of a psychiatric or physical (e.g., infectious disease) illness.
6. Inability to comply with restrictions and prohibited activities/treatments as listed in Section 3.3 of the Protocol.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (48):
  - University of Alabama at Birmingham - Division of Pulmonary, Allergy & Criticial Care, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center - Heart Lung Institute/ Clinical Research, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, Section of Pulmonary & Critical Care, New Haven, Connecticut
  - Advanced Pulmonary & Sleep Research Institute of Florida, Daytona Beach, Florida
  - University of Florida, Gainesville, Florida
  - ILD Research Center, Miami, Florida
  - Cleveland Clinic Florida- Weston Hospital, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - Via Christi Clinic, Wichita, Kansas
  - University of Kentucky- Center for Clinical and Translational Science, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Pulmonary Clinical Research Unit, Rochester, Minnesota
  - CardioPulmonary Research Center, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Pulmonary & Allergy Associates, PA, Summit, New Jersey
  - ISA Clinical Research, Forest Hills, New York
  - Weill Cornell Medical College, New York, New York
  - Highland Hospital, Rochester, New York
  - Asheville Pulmonary and Critical Care Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Pulmonary, Critical Care & Sleep Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Simmons Center for Interstitial Lung Disease, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Alamo Clinical Research, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Australia (5):
  - Local institution, Westmead, New South Wales
  - Local institution, Greenslopes, Queensland
  - Local Institution, Adelaide, South Australia
  - Local institution, Frankston, Victoria
  - Local institution, Nedlands, Western Australia
- Chile (4):
  - Local institution, Viña del Mar, Región de Valparaíso
  - Local institution, Quillota
  - Local institution, Santiago
  - Local Institution, Talca
- Colombia (4):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Fundacion Neumologica Colombiana, Bogota, Cundinamarca
  - Hospital Universitario San Ignacio, Bogota, Cundinamarca
  - Local Institution, Bogota, Cundinamarca
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Peru (2):
  - Local institution, Lima
  - Local Institution, Lima

REFERENCES:
- [Derived] Decato BE, Leeming DJ, Sand JMB, Fischer A, Du S, Palmer SM, Karsdal M, Luo Y, Minnich A. LPA1 antagonist BMS-986020 changes collagen dynamics and exerts antifibrotic effects in vitro and in patients with idiopathic pulmonary fibrosis. Respir Res. 2022 Mar 18;23(1):61. doi: 10.1186/s12931-022-01980-4. PMID 35303880
- [Derived] Palmer SM, Snyder L, Todd JL, Soule B, Christian R, Anstrom K, Luo Y, Gagnon R, Rosen G. Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial of BMS-986020, a Lysophosphatidic Acid Receptor Antagonist for the Treatment of Idiopathic Pulmonary Fibrosis. Chest. 2018 Nov;154(5):1061-1069. doi: 10.1016/j.chest.2018.08.1058. Epub 2018 Sep 7. PMID 30201408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 325 participants were enrolled,out of which 143 participants were randomized and treated. Reasons for not being treated were:Screening HRCT or Pulmonary function tests did not meet study criteria and "Other" reasons
Groups:
- BMS-986020 600 mg Once Daily: Participants received a dose of BMS-986020 300 milligram (mg) as oral tablets (each tablet of 300 mg*2) once daily (QD), for 26 weeks.
- BMS-986020 600 mg Twice Daily: Participants received a dose of BMS-986020 300 mg as oral tablets (each tablet of 300 mg*2) twice daily (BID), for 26 weeks.
- Placebo: Participants received placebo matched with BMS-986020 as oral tablets either QD or BID for 26 weeks.
Period: Overall Study
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Started | 48 | 48 | 47
Completed | 37 | 37 | 34
Not Completed | 11 | 11 | 13
Not completed — Drug-related adverse event | 1 | 2 | 1
Not completed — Drug-unrelated adverse event | 3 | 3 | 3
Not completed — Death | 1 | 1 | 0
Not completed — Unable to take study drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3
Not completed — Subject non-compliance | 0 | 1 | 2
Not completed — Physician Decision | 3 | 3 | 4
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo | Total
Number analyzed (Participants) | 48 | 48 | 47 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (6.53) | 69.1 (8.35) | 69.3 (7.57) | 68.9 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 14 | 41
  Male | 33 | 36 | 33 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 21 | 25 | 70
  Not Hispanic or Latino | 24 | 27 | 22 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 2 | 10
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 34 | 37 | 30 | 101
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 8 | 5 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Rate to Week 26
Description: FVC is the is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry; and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which is used to dilate participant's bronchial (breathing) tubes.
Time Frame: Baseline, Week 26
Population: Intent-to-treat (ITT) population included all randomized participants. Here 'N' 'number of participants analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 42 | 43 | 40
liters (L) | -0.076 (0.2238) | -0.050 (0.2440) | -0.136 (0.1804)

2. Secondary Outcome: Geometric Mean Ratio (GMR) of Quantitative Lung Fibrosis (QLF) Score at Week 26 to Baseline
Description: The QLF score itself ranges from 0 to 100%, where greater values represent a greater amount of lung fibrosis and are considered a worse health status. Hence smaller geometric mean ratios to baseline were considered favorable. Baseline included all testing done on Day -1 as well as predose on Day 1.
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants. Here 'N' 'number of participants analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Ratio
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 41 | 44 | 39
Ratio | 1.14 | 1.09 | 1.11

3. Secondary Outcome: Mean Change From Baseline in Six-minute Walk Test (6MWT) Distance to Week 26
Description: The 6MWT measures the distance (in meters), a participant is able to walk in 6 minutes. This test measures the distance a person can walk quickly on a flat, hard surface in 6 minutes and reflects an individual's ability to perform daily physical activities. Baseline included all testing done on Day -1 as well as predose on Day 1
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 42 | 43 | 40
meters (m) | -14.2 (47.85) | 6.1 (53.87) | 10.3 (54.73)

4. Secondary Outcome: Mean Change From Baseline in the University of California at San Diego Shortness of Breath Questionnaire (UCSD SOBQ) Total Score as a Measure of Dyspnea to Week 26
Description: The UCSD SOBQ is a 24-item questionnaire developed to measure breathlessness on a scale between zero and five where 0 is not at all breathless and 5 is maximally breathless or too breathless to do the activity. Baseline included all testing done on Day -1 as well as predose on Day 1. The total score ranges from 0 to 120, with higher scores indicating worse dyspnea.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 41 | 43 | 40
Unit on a scale | 3.8 (17.84) | -1.7 (21.29) | 3.9 (18.24)

5. Secondary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC) to Week 26
Description: FVC is is the total amount of air exhaled during the forced expiratory volume test that is measured during spirometry; and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of lungs after taking an inhaled bronchodilator medicine which is used to dilate bronchial (breathing) tubes. Baseline included all testing done on Day -1 as well as predose on Day 1
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 42 | 43 | 40
liters | -0.076 (0.2238) | -0.050 (0.2440) | -0.136 (0.1804)

6. Secondary Outcome: Mean Change From Baseline in Quality of Life as Measured by the Medical Outcomes Study (MOS) 36-Item Short-Form Health Survey (SF-36) to Week 26
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the Aggregate Physical score of the SF-36. Items 5-8 primarily contribute to the Aggregate mental score of the SF-36. Scores on each item are summed and averaged. Range for Aggregate Physical Score : 0=worst to 100=best; and for Aggregate Mental Score: 0=worst to 100=best. Increases from baseline indicate improvement. Baseline included all testing done on Day -1 as well as predose on Day 1
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants. Here 'N' 'number of participants analyzed' signifies number of participants who were evaluable for each category.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 41 | 43 | 40
Units on a scale
  Aggregate Physical Score | -3.4 (1.0) | -1.0 (1.0) | -2.1 (1.1)
  Aggregate Mental Score | 0.1 (1.3) | 1.7 (1.3) | -1.1 (1.3)

7. Secondary Outcome: Number of Participants With Death or Non-Elective Hospitalization
Description: Time to death or non-elective hospitalization was defined as the elapsed time (days) from randomization to the date of death or the first non-elective hospitalization.
Time Frame: Upto Day 210
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 48 | 48 | 47
Participants | 5 | 4 | 2

8. Secondary Outcome: Number of Participants With Death or Respiratory Hospitalization or 10 Percent (%) Decline in Absolute Volume of FVC or 25-Meter Loss in 6-Minute Walk Distance (6MWD)
Description: Number of participants with death or respiratory hospitalization or 10% decline in absolute volume of FVC or 25 meter loss in 6MWD over time were reported.
Time Frame: Upto Day 210
Population: Safety Population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 48 | 48 | 47
Participants | 24 | 28 | 26

9. Secondary Outcome: Mean Change From Baseline in Carbon Monoxide Diffusing Capacity (DLCO) to Week 26
Description: DLCO is a measurement of the ability of the lungs to transfer gases from the air to the blood. Participant breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participant hold the breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine how much of the tracer gas was absorbed during the breath. DLCO, both uncorrected and corrected for hemoglobin in milliliter per minute per millimeter of mercury (mL/min/mmHg) was assessed.
Time Frame: Baseline, Week 26
Population: ITT population included all randomized participants.Here 'n' 'number analyzed' signifies number of participants who were evaluable for each category.
Measure: Least Squares Mean (Standard Error); unit: mL/min/mmHg
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 40 | 43 | 39
mL/min/mmHg
  Uncorrected for hemoglobin | -1.1 (0.7) | -0.2 (0.7) | -1.1 (0.7)
  Corrected for hemoglobin | -1.2 (0.7) | -0.2 (0.7) | -1.1 (0.7)

10. Secondary Outcome: Number of Participants With Definite or Probable Acute Exacerbation (AEx) of Idiopathic Pulmonary Fibrosis (IPF)
Description: Acute IPF exacerbations is defined as a clinically significant deterioration of unidentifiable cause in a participant with underlying IPF. Exacerbations of IPF were adjudicated as definite (>=1 AEx) and Probable. Investigators were asked to make the diagnosis of acute exacerbation of IPF on the basis of subjective worsening over 30 days or less, new bilateral radiographic opacities, and the absence of infection or another identifiable etiology. The final diagnosis, however, was confirmed by the study medical monitor.
Time Frame: Upto Day 210
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
Number analyzed (Participants) | 48 | 48 | 47
Participants
  Definite | 0 | 2 | 0
  Probable | 1 | 1 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) BMS-986020
Description: Cmax is defined as the maximum observed plasma concentration.
Time Frame: Day 1 and Day 7
Population: Evaluable pharamcokinetic (PK) population included all participants who have adequate PK profiles. Here 'n' 'number analyzed' signifies number of participants evaluable at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (ug/L)
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
microgram per liter (ug/L)
  Day 1 | 5963.7 (65) | 3005.8 (104)
  Day 7: number analyzed (Participants) | 5 | 7
  Day 7 | 6535.4 (68) | 7266.2 (51)

12. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of BMS-986020
Description: Tmax is defined as the maximum observed plasma concentration.
Time Frame: Day 1 and Day 7
Population: Evaluable PK population included all participants who have adequate PK profiles. Here 'n' 'number analyzed' signifies number of participants evaluable at each time point.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
hours (h)
  Day 1 | 3.110 [1.07 to 6.00] | 2.030 [1.00 to 4.00]
  Day 7: number analyzed (Participants) | 5 | 7
  Day 7 | 3.000 [1.02 to 4.00] | 2.000 [0.50 to 3.00]

13. Secondary Outcome: Accumulation Index (AI) of BMS-986020
Description: AI is the ratio of area under the concentration time curve in one dosing interval in (AUC[TAU]) at steady-state to AUC(TAU) after the first dose.
Time Frame: Day 7
Population: Evaluable PK population included all participants who have adequate PK profiles. Here 'n' 'number analyzed' signifies number of participants evaluable this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 5 | 7
Ratio | 1.2329 (80) | 1.9386 (97)

14. Secondary Outcome: Area Under the Concentration Time Curve in One Dosing Interval of BMS -986020 in at Steady-state
Description: AUC(TAU) is the area under the concentration time curve in one dosing interval in at steady-state.
Time Frame: Day 1 and Day 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/L
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
ug*h/L
  Day 1 | 26921.6 (69) | 11689.5 (83)
  Day 7: number analyzed (Participants) | 5 | 7
  Day 7 | 29174.1 (46) | 22661.8 (51)

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over 12 Hours Post-dose AUC(0-12) of BMS -986020
Description: AUC(0-12) is the area under the plasma concentration time curve over 12 hours post-dose.
Time Frame: Day 1 and Day 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/L
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
ug*h/L
  Day 1 | 21014.1 (60) | 11689.5 (83)
  Day 7: number analyzed (Participants) | 5 | 7
  Day 7 | 24242.3 (51) | 22661.8 (51)

16. Secondary Outcome: Apparent Oral Clearance (CLF/F) of BMS -986020
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 1 and Day 7
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
Liter per hour (L/h)
  Day 1 | 20.272 (79) | 43.846 (94)
  Day 7: number analyzed (Participants) | 5 | 7
  Day 7 | 20.566 (41) | 26.476 (60)

17. Secondary Outcome: Average Concentration of BMS -986020 at Steady State (Css[Avg])
Description: Css (avg) is the average concentration at steady state.
Time Frame: Day 7
Population: Evaluable PK population included all participants who have adequate PK profiles. Here 'n' 'number analyzed' signifies number of participants evaluable at this time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/L
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily
Number analyzed (Participants) | 6 | 7
ug/L | 1215.6 (46) | 1888.5 (51)

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from signature of the informed consent until 4 weeks after last treatment administration
Description: Analysis was performed on safety population which included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | BMS-986020 600 mg Once Daily | BMS-986020 600 mg Twice Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 2/48 | 2/48 | 1/47
Serious Adverse Events (participants affected / at risk) | 9/48 | 16/48 | 12/47
Other Adverse Events (participants affected / at risk) | 21/48 | 40/48 | 25/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-986020 600 mg Once Daily (N=48) | BMS-986020 600 mg Twice Daily (N=48) | Placebo (N=47)
Overdose (Injury, poisoning and procedural complications) | 1 | 4 | 6
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986020 600 mg Once Daily (N=48) | BMS-986020 600 mg Twice Daily (N=48) | Placebo (N=47)
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 5 | 0
Bronchitis (Infections and infestations) | 6 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Fatigue (General disorders) | 4 | 8 | 2
Gastritis (Gastrointestinal disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 2 | 8 | 4
Hepatic enzyme increased (Investigations) | 0 | 4 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Nasopharyngitis (Infections and infestations) | 5 | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 2 | 2
Pharyngitis (Infections and infestations) | 3 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 3
Transaminases increased (Investigations) | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5

LIMITATIONS AND CAVEATS:
Due to 3 SAE cases on active treatment, a decision was taken by the sponsor to immediately discontinue all study dosing and to implement additional post-treatment safety monitoring in the off-treatment follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.